CLINICAL TRIAL: NCT04531384
Title: Randomized Clinical Trial of Robot-Assisted Intelligent Rehabilitation Treatment in Comparison With Standard Treatment for Methamphetamine Use Disorders and Alcohol Use Disorders
Brief Title: Robot-Assisted Intelligent Rehabilitation Treatment for Methamphetamine Use Disorders.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MZhao-010
Record Dates: First submitted 2020-08-04; First posted 2020-08-28 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-09

CONDITIONS: Amphetamine Addiction
MeSH Terms: conditions — Amphetamine-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robot-assisted rehabilitation intelligent treatment (Experimental): Participants assigned to this condition were offered 10 weekly individual sessions of robot-assisted rehabilitation treatment, delivered by the Robot-assisted rehabilitation intelligent system. The system contains 10 core cognitive-behavioral therapy (CBT) skill topics (such as functional analysis, coping skills training, reviewing practice exercises, explaining CBT concepts). A robot therapist demonstrates the target CBT skills and assigns homework to participants.
  Interventions: Device: robot-assisted rehabilitation intelligent treatment
- treatment as usual (Other): Participants in the treatment-as-usual group were offered standard treatment at the compulsory isolated detoxification centers and non-compulsory isolated detoxification institutions, which consisted of weekly group and/or individual therapy, as determined by the clinical team.
  Interventions: Other: standard psychotherapy treatment

INTERVENTIONS:
Device: robot-assisted rehabilitation intelligent treatment — robot-assisted rehabilitation psychotherapy
  Arms: robot-assisted rehabilitation intelligent treatment
Other: standard psychotherapy treatment — standard treatment at the compulsory isolated detoxification centers and non-compulsory isolated detoxification institutions
  Arms: treatment as usual

SUMMARY:
The purpose of this research is to evaluate the efficacy and safety of Robot-assisted rehabilitation intelligent system as a virtual stand-alone treatment, delivered with minimal clinical monitoring compared with treatment as usual in methamphetamine (MA) use disorders.

DETAILED DESCRIPTION:
Based on artificial intelligence technology, face recognition technology, virtual reality technology to develop an available Robot-assisted rehabilitation intelligent system. Then, using this intelligent system as a new way of Psychotherapy to provide treatment for methamphetamine patients, and compare it with traditional treatment to verify the efficacy and safety of Robot-assisted rehabilitation intelligent system in Chinese methamphetamine patients.

ELIGIBILITY:
Inclusion Criteria:

* In accordance with the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) for methamphetamine (MA) use disorders;
* Education level equal or more than 9 years;
* Have normal or corrected-to-normal vision;
* Have normal or corrected-to-normal hearing;
* Less than 3 months before last drug use;

Exclusion Criteria:

* Current substance use (except nicotine or caffeine);
* History of disease which influence cognition，such as seizure disorder、cerebrovascular disease、head injury or other severe medication conditions;
* Intelligence quotient less than 70.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Changes of galvanic skin response during the virtual reality based addiction assessment system | in 1 year
  The galvanic skin response is an emotional physiological indicator, and its unit is ohm.

SECONDARY OUTCOMES:
Treatment motivation | in 1 year
  Using the Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES) to measure the treatment motivation of the participants. The score of the scale is between 19 and 95. The higher the score, the higher the treatment motivation.
Anxiety | in 1 year
  Anxiety is assessed by the State-Trait Anxiety Scale (SAS). The score of the SAS scale is between 0 and 80. The higher the score, the more severe the anxiety symptoms.
Depression | in 1 year
  Depression is assessed by the the Beck Depression Scale (SDS). The score of the SDS scale is between 0 and 80. The higher the score, the more severe the depression symptoms.
Attentional bias related to drugs and emotional stimulation | in 1 year
  The emotional Stroop tests is used for assessed attentional bias. The indicator is the accuracy rate of the key presses, from 0 to 100%.
Risky decision-making | in 1 year
  Balloon Analogue Risk Task is used for assess the risky decision-making ability. The indicator is the average number of balloon blows, and its unit is times.
Reaction inhibition ability | in 1 year
  Stop signal task is used for assess the reaction inhibition ability. The indicator is the reaction time when the participant completes the task, and its unit is milliseconds.
Changes of electroencephalogram power spectrum during the virtual reality based addiction | in 1 year
  The electroencephalogram power spectrum reflects the functional status of the brain, and its unit is uV^2.

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhao, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Gaojing Rehabilitation Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No